CLINICAL TRIAL: NCT02461875
Title: Cabergoline Versus GnRH Antagonist Rescue and Cabergoline in the Prevention of Ovarian Hyperstimulation Syndrome: a Randomized Controlled Trial
Brief Title: Cabergoline Versus GnRH Antagonist Rescue and Cabergoline in the Prevention of Ovarian Hyperstimulation Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Prof .Usama M.Fouda, M.D , PhD, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cabergoline / GnRH antagonist
Record Dates: First submitted 2015-05-29; First posted 2015-06-03 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: OHSS
Keywords: OHSS; Infertility; Cabergoline; GnRH antagonist; IVF-ET
MeSH Terms: conditions — Infertility | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabergoline group (Active Comparator): Cabergoline is administered starting on the day of HCG administration.
  Interventions: Drug: Cabergoline
- GnRH antagonist rescue & cabergoline group (Experimental): Converting a long GnRH agonist cycle to an GnRH antagonist cycle (GnRH antagonist rescue) and Cabergoline is administered starting on the day of HCG administration.
  Interventions: Drug: GnRH antagonist rescue & cabergoline

INTERVENTIONS:
Drug: Cabergoline — Patients receive cabergoline 0.5 mg p.o at bed time for 8 days starting on the day of HCG administration.
  Arms: Cabergoline group
Drug: GnRH antagonist rescue & cabergoline — when the leading follicle reaches 16 mm, HP-uFSH is continued at daily dose of 75 IU/day till the day of HCG administration. Moreover, Gn RH agonist (triptorelin) is discontinued and GnRH antagonist (Cetrorelix acetate)0.25 mg S.C is administered daily till the day of HCG administration. Serum estradiol is measured daily and HCG (5,000 IU/I.M) is administered when serum estradiol level drops below 3500 pg/ml . Moreover, cabergoline 0.5 mg p.o is administered at bed time for 8 days starting on the day of HCG administration.
  Arms: GnRH antagonist rescue & cabergoline group

SUMMARY:
The aim of study is to compare the efficacy of GnRH antagonist rescue combined with cabergoline with cabergoline in the prevention of ovarian hyperstimulation syndrome in high risk patients undergoing ovarian stimulation for IVF-ET with long GnRH agonist protocol.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is the most serious complication of assisted reproduction. Complications of OHSS include vascular thrombosis, pulmonary embolism, renal failure, electrolyte disturbances, ascites, hydrothorax ,torsion of the ovary, abortion or rarely death.

Previous studies revealed that converting a long GnRH agonist cycle to an GnRH antagonist cycle (GnRH antagonist rescue) reduced the risk of OHSS. Other studies revealed that cabergoline (potent dopamine receptor agonist on D2 receptors)was effective in preventing OHSS.

The aim of study is to compare the efficacy of GnRH antagonist rescue combined with cabergoline with cabergoline in the prevention of ovarian hyperstimulation syndrome in high risk patients undergoing ovarian stimulation for IVF-ET with long GnRH agonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ovarian stimulation for IVF-ET with long GnRH agonist protocol and at high risk of developing OHSS [ have more than 20 follicles ( 90% of them less than 14 mm in mean diameter) and serum estradiol ≥ 3000 pg/ml]

Exclusion Criteria:

* Fibrosis of lung,
* swelling or inflammation around the heart or lung,
* hypertension,
* liver disease,
* heart valve disease and
* allergy to cabergoline or ergot derivatives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Moderate or severe ovarian hyperstimulation syndrome | Within 4 weeks of HCG adminstration

SECONDARY OUTCOMES:
The Number of Participants Who Achieved Ongoing Pregnancy | 18 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Chair — Aljazeera (Al Gazeera) hospital
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Giza Governorate, Egypt

REFERENCES:
- [Background] Aboulghar MA, Mansour RT, Amin YM, Al-Inany HG, Aboulghar MM, Serour GI. A prospective randomized study comparing coasting with GnRH antagonist administration in patients at risk for severe OHSS. Reprod Biomed Online. 2007 Sep;15(3):271-9. doi: 10.1016/s1472-6483(10)60339-2. PMID 17854523
- [Derived] Fouda UM, Sayed AM, Elshaer HS, Hammad BE, Shaban MM, Elsetohy KA, Youssef MA. GnRH antagonist rescue protocol combined with cabergoline versus cabergoline alone in the prevention of ovarian hyperstimulation syndrome: a randomized controlled trial. J Ovarian Res. 2016 May 17;9(1):29. doi: 10.1186/s13048-016-0237-8. PMID 27184139